CLINICAL TRIAL: NCT02907424
Title: Comparison of a Locally Produced RUTF With a Commercial RUTF in the Treatment of SAM in Cambodia
Brief Title: Comparison of a Locally Produced RUTF With a Commercial RUTF in the Treatment of SAM
Acronym: FLNS_SAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ministry of Agriculture, Forestry and Fisheries Cambodia (Unknown); UNICEF (Other)
Responsible Party: Principal Investigator, Frank Wieringa, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRD_UNICEF_DFPTQ_SAM
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition; Children; Treatment
MeSH Terms: conditions — Malnutrition | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BP-100 (Active Comparator): standard treatment
  Interventions: Dietary Supplement: 2 months of treatment
- Num Trey (Experimental): locally produced RUTF
  Interventions: Dietary Supplement: 2 months of treatment

INTERVENTIONS:
Dietary Supplement: 2 months of treatment — standard 2 months of treatment

SUMMARY:
In order to make Cambodia independent from importing a product for the treatment and prevention of malnutrition, UNICEF, DFPTQ Fisheries Administration and IRD have started a collaboration for the development of a range of products for the treatment and prevention of malnutrition. To reduce costs of the product, and to adapt the taste to local circumstances, the protein source of the usual RUTF (milk powder) has been changed to fish (Trey Riel). The main objective of this sub-study is to test the efficacy of the newly developed RUTF on the recovery of children suffering from severe acute malnutrition. As comparison, the current treatment of SAM with BP-100 will be used.

ELIGIBILITY:
Inclusion Criteria:

* discharged from hospital after admission for SAM
* WHZ <2.8 Z-score or MUAC<11.5 cm
* no complications
* passing the appetite test

Exclusion Criteria:

* <6 mo of age
* complications related to SAM

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
weight gain | 2 months
  weight gain in g/kg/day

SECONDARY OUTCOMES:
body composition | 2 months
  changes in body composition obtained from skinfold thickness measurements over the treatment period
Fatty Acid composition | 2 months
  changes in serum concentrations of fatty acids over the intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Fisheries Post-harvest Technologies and Quality Control, Fisheries Administration, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sigh S, Lauritzen L, Wieringa FT, Laillou A, Chamnan C, Stark KD, Roos N. Changes in polyunsaturated fatty acids during treatment of malnourished children may be insufficient to reach required essential fatty acid levels - A randomised controlled trial. Clin Nutr. 2023 Sep;42(9):1778-1787. doi: 10.1016/j.clnu.2023.08.003. Epub 2023 Aug 6. PMID 37572581
- [Derived] Sigh S, Lauritzen L, Wieringa FT, Laillou A, Chamnan C, Angkeabos N, Moniboth D, Berger J, Stark KD, Roos N. Whole-blood PUFA and associations with markers of nutritional and health status in acutely malnourished children in Cambodia. Public Health Nutr. 2020 Apr;23(6):974-986. doi: 10.1017/S1368980019003744. Epub 2020 Jan 24. PMID 31973779